CLINICAL TRIAL: NCT04356404
Title: Risk of Hepatitis Flare in Patients With Previous Hepatitis B Virus Exposure Amongst Patients on Immunosuppressive and Biological Modifier Therapies Exposure
Brief Title: Risk of Hepatitis Flare in Patients With Previous Hepatitis B Virus Exposure Amongst Patients
Status: Terminated | Type: Observational
Why Stopped: No suitable case identified
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Principal Investigator, Mak Wing Yan, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: HEP-FLARE_Protocol_20210604_V5
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Occult Hepatitis B; Biological Substance; Adverse Effect; Immunosuppression
Keywords: Occult Hepatitis B infection; Biologics; Immunosuppressants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective group: Patients will be followed up until development of hepatitis flare or at 2 years after study recruitment. We plan to recruit 150 patients for the prospective cohort.

SUMMARY:
The purpose of this study is to study the risk of hepatitis flare in patients with previous hepatitis B virus exposure amongst patients on immunosuppressive and biological modifier therapies

DETAILED DESCRIPTION:
Chronic hepatitis B infection remains a global health threat despite vaccination program.[1] Nearly 3 billion population are infected with chronic hepatitis B infection globally. In China, the pooled prevalence of chronic hepatitis B infection was around 7% in year 2018, making an estimated 84 millions of population living with chronic hepatitis B infection. Hepatitis B virus infection is the leading cause of liver cirrhosis and hepatocellular carcinoma, leading to significant morbidity and mortality. Patients with hepatitis B infection can present with a wide range of clinical presentation, ranging from inactive carrier to fulminant hepatitis, cirrhosis or development of hepatocellular carcinoma. Besides, a significant proportion of patients are suffering from occult hepatitis B infection (OBI), which is defined as a state of undetectable serum HBsAg yet detectable serum and/ or intrahepatic HBV DNA. Report from the European Association for the Study of the Liver (EASL) in 2008 has revealed that around one-third of the global population has serological evidence of past or present HBV infection. Disappearance of HBsAg, also known as HBsAg seroclearance, can occur either spontaneously or after anti-viral treatment. However, patients with past or resolved HBV infection are still at risk of development of hepatocellular carcinoma, liver cirrhosis and liver-related mortality.The reported prevalence of OBI amongst patients with non-alcoholic fatty liver disease in Hong Kong was 35% (submitted to American Journal of Gastroenterology, under review). It is well known that there is risk of HBV reactivation after chemotherapy or immunosuppressive therapy which can lead to fulminant liver failure or even death. Short course of high dose corticosteroid could increase the risk of hepatitis flare in patients with chronic hepatitis B infection. Even in patients with OBI, a high daily dose of corticosteroid (>40mg prednisolone equivalents) increased risks of hepatitis flare. It is thus important to know the hepatitis B virus status before start of chemotherapy, immunosuppressive therapy or corticosteroid.

Biologics is one of the mainstay treatments for many autoimmune diseases, including inflammatory bowel disease (IBD), rheumatoid arthritis (RA) and systemic lupus erythematosus (SLE), psoriasis etc. The incidence of IBD has increased rapidly in Hong Kong over the past 30 years. The age-adjusted incidence of IBD in Hong Kong has rose from 0.10 per 100,000 individuals in 1985 to 3.12 per 100,000 individuals in 2014. The reported prevalence of RA in Hong Kong was 0.35% while the reported prevalence of SLE in Hong Kong was 0.1% with annual incidence of 6.7 per 100,000 individuals. It is well known that treatment with biological agent like anti-CD20 monoclonal antibody (rituximab) in patients with OBI can lead to fulminant hepatitis B flare. Recently, anti-tumor necrosis factor alpha (TNF α) has been widely used in patients with inflammatory bowel disease and various rheumatological diseases. Risk of hepatitis B reactivation after anti-TNF α has been reported, but actual risk remains controversial. In a report from Japan including 135 rheumatoid arthritis patients with previous HBV infections, 17/135 (12.6%) had HBV reactivation after receiving immunosuppressants and patients who were treated with biologics were more frequent to develop HBV reactivation compared to those who were not on biologics. In another study, 9/168 (5%) anti-HBc positive patients developed HBV reactivation after receiving anti-TNF α and one patient died due to fulminant liver failure.However, another three studies revealed low rates of HBV reactivation (0-2%) amongst rheumatology patients with previous HBV infections receiving anti-TNF α. The European Crohn's and Colitis Organisation (ECCO) suggested routine antiviral prophylaxis for patients with previous HBV infection starting biologics is not recommended. Instead, regular monitoring of ALT/ AST, change in HBV serology and HBV DNA every 1 to 3 months should be performed. In 2015, the American Gastroenterology Association (AGA) has developed guideline on the prevention and treatment of hepatitis B virus reactivation during immunosuppressive therapy. It classifies patients receiving anti-TNF α as moderate risk of developing HBV reactivation and antiviral prophylaxis is preferred over monitoring alone, but it is a weak recommendation. Therefore, it is now still uncertain whether prophylactic anti-viral should be given for patients with previous HBV exposure before starting anti-TNF α.

With the advancement of technology, there are now more biological agents and small molecules for the treatment of IBD and various rheumatological conditions. These include anti-integrin, cytokine inhibitors, and small molecules e.g. JAK inhibitors. Cytokine inhibitor, ustekinumab (anti-IL12/23), has been reported to be leading to hepatitis reactivation in a psoriasis patient who has past HBV infection.[26] Whether these agents can lead to hepatitis flare in patients with past HBV exposure remains largely unknown.

Based on the compelling data, the investigators hypothesize that use of biologic modifier therapies in patients with occult hepatitis B infection will lead to hepatitis flare. The investigators aim to assess the rate of hepatitis flare while on biological modifier therapies in both retrospective population-based database and prospectively in patients who are on biological modifier therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at the time of starting biological modifier therapies or at the time of recruitment
* Positive for anti-HBc OR
* Positive for anti-HBs and born before year 1988

Exclusion Criteria:

* Known HBV carrier with HBsAg positive
* Concomitant HCV and/ or HIV infection
* Already on HBV anti-viral
* Refuse to consent
* Baseline ALT > 80 IU/ml

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with previous HBV exposure who are already on biological modifier therapies and who will be newly started on biological modifier therapies in the Department of Medicine and Therapeutics, Prince of Wales Hospital and Department of Medicine, University Malaya Medical Centre will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Rate of hepatitis flare | 24 months
  Hepatitis flare, defined as ALT >2xULN IU/L, according to the Asia Pacific Association for the Study of the Liver (APASL) definition while on biological modifier therapy. The upper limit of normal (ULN) was defined as 40 IU/L by APASL.

SECONDARY OUTCOMES:
Rate of severe hepatitis flare | 24 months
  Severe hepatitis flare, defined as ALT > 5xULN or > 10xULN, as defined by the APASL definition, while on biological modifier therapy
Rate of icteric flare | 24 months
  Icteric flare, defined as ALT raised >3xULN together with serum total bilirubin >2xULN (i.e. >38 µmol/L), while on biological modifier therapy
Rate of HBsAg seroreversion | 24 months
  HBsAg seroreversion, defined as reappearance of HBsAg
Risk factors associated with development of hepatitis flare | 24 months
  Risk factors associated with development of hepatitis flare, Including concomitant use of steroid and immunosuppressants

CONTACTS AND LOCATIONS:
Overall Officials: WingYan Mak, MRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polaris Observatory Collaborators. Global prevalence, treatment, and prevention of hepatitis B virus infection in 2016: a modelling study. Lancet Gastroenterol Hepatol. 2018 Jun;3(6):383-403. doi: 10.1016/S2468-1253(18)30056-6. Epub 2018 Mar 27. PMID 29599078
- [Background] Wang H, Men P, Xiao Y, Gao P, Lv M, Yuan Q, Chen W, Bai S, Wu J. Hepatitis B infection in the general population of China: a systematic review and meta-analysis. BMC Infect Dis. 2019 Sep 18;19(1):811. doi: 10.1186/s12879-019-4428-y. PMID 31533643
- [Background] Maynard JE. Hepatitis B: global importance and need for control. Vaccine. 1990 Mar;8 Suppl:S18-20; discussion S21-3. doi: 10.1016/0264-410x(90)90209-5. PMID 2139281
- [Background] Torbenson M, Thomas DL. Occult hepatitis B. Lancet Infect Dis. 2002 Aug;2(8):479-86. doi: 10.1016/s1473-3099(02)00345-6. PMID 12150847
- [Background] Raimondo G, Allain JP, Brunetto MR, Buendia MA, Chen DS, Colombo M, Craxi A, Donato F, Ferrari C, Gaeta GB, Gerlich WH, Levrero M, Locarnini S, Michalak T, Mondelli MU, Pawlotsky JM, Pollicino T, Prati D, Puoti M, Samuel D, Shouval D, Smedile A, Squadrito G, Trepo C, Villa E, Will H, Zanetti AR, Zoulim F. Statements from the Taormina expert meeting on occult hepatitis B virus infection. J Hepatol. 2008 Oct;49(4):652-7. doi: 10.1016/j.jhep.2008.07.014. Epub 2008 Jul 31. No abstract available. PMID 18715666
- [Background] Yip TC, Chan HL, Wong VW, Tse YK, Lam KL, Wong GL. Impact of age and gender on risk of hepatocellular carcinoma after hepatitis B surface antigen seroclearance. J Hepatol. 2017 Nov;67(5):902-908. doi: 10.1016/j.jhep.2017.06.019. Epub 2017 Jun 24. PMID 28652084
- [Background] Yip TC, Wong GL, Chan HL, Tse YK, Lam KL, Lui GC, Wong VW. HBsAg seroclearance further reduces hepatocellular carcinoma risk after complete viral suppression with nucleos(t)ide analogues. J Hepatol. 2019 Mar;70(3):361-370. doi: 10.1016/j.jhep.2018.10.014. Epub 2018 Oct 25. PMID 30367899
- [Background] Yip TC, Wong GL, Wong VW, Tse YK, Lui GC, Lam KL, Chan HL. Durability of hepatitis B surface antigen seroclearance in untreated and nucleos(t)ide analogue-treated patients. J Hepatol. 2017 Oct 6:S0168-8278(17)32332-2. doi: 10.1016/j.jhep.2017.09.018. Online ahead of print. PMID 28989093
- [Background] Chung SM, Sohn JH, Kim TY, Yoo KD, Ahn YW, Bae JH, Jeon YC, Choi JH. [Fulminant hepatic failure with hepatitis B virus reactivation after rituximab treatment in a patient with resolved hepatitis B]. Korean J Gastroenterol. 2010 Apr;55(4):266-9. doi: 10.4166/kjg.2010.55.4.266. Korean. PMID 20389182
- [Background] Khan ZH, Ilyas K, Ghazanfar H, Khan HH, Hussain Q, Hammad S, Munir A, Asim R. Fatal Fulminant Hepatitis from Rituximab-induced Hepatitis B Reactivation in a Patient with Follicular Lymphoma: A Case Report and a Brief Review of Literature. Cureus. 2018 Mar 2;10(3):e2257. doi: 10.7759/cureus.2257. PMID 29725560
- [Background] Ng SC, Leung WK, Shi HY, Li MK, Leung CM, Ng CK, Lo FH, Hui YT, Tsang SW, Chan YK, Loo CK, Chan KH, Hui AJ, Chow WH, Harbord M, Ching JY, Lee M, Chan V, Tang W, Hung IF, Ho J, Lao WC, Wong MT, Sze SF, Shan EH, Lam BC, Tong RW, Mak LY, Wong SH, Wu JC, Chan FK, Sung JJ. Epidemiology of Inflammatory Bowel Disease from 1981 to 2014: Results from a Territory-Wide Population-Based Registry in Hong Kong. Inflamm Bowel Dis. 2016 Aug;22(8):1954-60. doi: 10.1097/MIB.0000000000000846. PMID 27416041
- [Background] Ho CTK, Mok CC, Cheung TT, Kwok KY, Yip RML; Hong Kong Society of Rheumatology. Management of rheumatoid arthritis: 2019 updated consensus recommendations from the Hong Kong Society of Rheumatology. Clin Rheumatol. 2019 Dec;38(12):3331-3350. doi: 10.1007/s10067-019-04761-5. Epub 2019 Sep 4. PMID 31485846
- [Background] Mok CC. Epidemiology and survival of systemic lupus erythematosus in Hong Kong Chinese. Lupus. 2011 Jun;20(7):767-71. doi: 10.1177/0961203310388447. Epub 2010 Dec 10. PMID 21148605
- [Background] Sera T, Hiasa Y, Michitaka K, Konishi I, Matsuura K, Tokumoto Y, Matsuura B, Kajiwara T, Masumoto T, Horiike N, Onji M. Anti-HBs-positive liver failure due to hepatitis B virus reactivation induced by rituximab. Intern Med. 2006;45(11):721-4. doi: 10.2169/internalmedicine.45.1590. Epub 2006 Jul 3. PMID 16819252
- [Background] Koo YX, Tay M, Teh YE, Teng D, Tan DS, Tan IB, Tai DW, Quek R, Tao M, Lim ST. Risk of hepatitis B virus (HBV) reactivation in hepatitis B surface antigen negative/hepatitis B core antibody positive patients receiving rituximab-containing combination chemotherapy without routine antiviral prophylaxis. Ann Hematol. 2011 Oct;90(10):1219-23. doi: 10.1007/s00277-011-1241-0. Epub 2011 Apr 26. PMID 21520001
- [Background] Urata Y, Uesato R, Tanaka D, Kowatari K, Nitobe T, Nakamura Y, Motomura S. Prevalence of reactivation of hepatitis B virus replication in rheumatoid arthritis patients. Mod Rheumatol. 2011 Feb;21(1):16-23. doi: 10.1007/s10165-010-0337-z. Epub 2010 Jul 29. PMID 20668905
- [Background] Perez-Alvarez R, Diaz-Lagares C, Garcia-Hernandez F, Lopez-Roses L, Brito-Zeron P, Perez-de-Lis M, Retamozo S, Bove A, Bosch X, Sanchez-Tapias JM, Forns X, Ramos-Casals M; BIOGEAS Study Group. Hepatitis B virus (HBV) reactivation in patients receiving tumor necrosis factor (TNF)-targeted therapy: analysis of 257 cases. Medicine (Baltimore). 2011 Nov;90(6):359-371. doi: 10.1097/MD.0b013e3182380a76. PMID 22033451
- [Background] Caporali R, Bobbio-Pallavicini F, Atzeni F, Sakellariou G, Caprioli M, Montecucco C, Sarzi-Puttini P. Safety of tumor necrosis factor alpha blockers in hepatitis B virus occult carriers (hepatitis B surface antigen negative/anti-hepatitis B core antigen positive) with rheumatic diseases. Arthritis Care Res (Hoboken). 2010 Jun;62(6):749-54. doi: 10.1002/acr.20130. PMID 20535784
- [Background] Tamori A, Koike T, Goto H, Wakitani S, Tada M, Morikawa H, Enomoto M, Inaba M, Nakatani T, Hino M, Kawada N. Prospective study of reactivation of hepatitis B virus in patients with rheumatoid arthritis who received immunosuppressive therapy: evaluation of both HBsAg-positive and HBsAg-negative cohorts. J Gastroenterol. 2011 Apr;46(4):556-64. doi: 10.1007/s00535-010-0367-5. Epub 2011 Jan 19. PMID 21246383
- [Background] Lee YH, Bae SC, Song GG. Hepatitis B virus (HBV) reactivation in rheumatic patients with hepatitis core antigen (HBV occult carriers) undergoing anti-tumor necrosis factor therapy. Clin Exp Rheumatol. 2013 Jan-Feb;31(1):118-21. Epub 2012 Oct 30. PMID 23111095
- [Background] Rahier JF, Magro F, Abreu C, Armuzzi A, Ben-Horin S, Chowers Y, Cottone M, de Ridder L, Doherty G, Ehehalt R, Esteve M, Katsanos K, Lees CW, Macmahon E, Moreels T, Reinisch W, Tilg H, Tremblay L, Veereman-Wauters G, Viget N, Yazdanpanah Y, Eliakim R, Colombel JF; European Crohn's and Colitis Organisation (ECCO). Second European evidence-based consensus on the prevention, diagnosis and management of opportunistic infections in inflammatory bowel disease. J Crohns Colitis. 2014 Jun;8(6):443-68. doi: 10.1016/j.crohns.2013.12.013. Epub 2014 Mar 6. No abstract available. PMID 24613021
- [Background] Reddy KR, Beavers KL, Hammond SP, Lim JK, Falck-Ytter YT; American Gastroenterological Association Institute. American Gastroenterological Association Institute guideline on the prevention and treatment of hepatitis B virus reactivation during immunosuppressive drug therapy. Gastroenterology. 2015 Jan;148(1):215-9; quiz e16-7. doi: 10.1053/j.gastro.2014.10.039. Epub 2014 Oct 31. No abstract available. PMID 25447850
- [Background] Koskinas J, Tampaki M, Doumba PP, Rallis E. Hepatitis B virus reactivation during therapy with ustekinumab for psoriasis in a hepatitis B surface-antigen-negative anti-HBs-positive patient. Br J Dermatol. 2013 Mar;168(3):679-80. doi: 10.1111/bjd.12120. Epub 2013 Jan 31. No abstract available. PMID 23121260
- [Background] Wong GL, Wong VW, Yuen BW, Tse YK, Yip TC, Luk HW, Lui GC, Chan HL. Risk of hepatitis B surface antigen seroreversion after corticosteroid treatment in patients with previous hepatitis B virus exposure. J Hepatol. 2020 Jan;72(1):57-66. doi: 10.1016/j.jhep.2019.08.023. Epub 2019 Sep 6. PMID 31499132
- [Background] Wong GL, Yuen BW, Chan HL, Tse YK, Yip TC, Lam KL, Lui GC, Wong VW. Impact of dose and duration of corticosteroid on the risk of hepatitis flare in patients with chronic hepatitis B. Liver Int. 2019 Feb;39(2):271-279. doi: 10.1111/liv.13953. Epub 2018 Sep 25. PMID 30179316
- [Background] Yip TC, Wong GL. Current Knowledge of Occult Hepatitis B Infection and Clinical Implications. Semin Liver Dis. 2019 May;39(2):249-260. doi: 10.1055/s-0039-1678728. Epub 2019 Mar 25. PMID 30912100